CLINICAL TRIAL: NCT05242172
Title: THE RELATIONSHIP OF CRP/ALBUMIN RATIO LEVEL AND PROGNOSIS IN PREGNANT COVID-19 PATIENTS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Nezir Yılmaz, Principal investigator, Adiyaman University Research Hospital
Other Study IDs: 14/12/2021-2021/10-19
Record Dates: First submitted 2022-02-15; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-01

CONDITIONS: Corona Virus Infection; Pregnancy; Infection
MeSH Terms: conditions — Coronavirus Infections; Pregnancy Complications, Infectious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CRP/Albumin ratio — it is aimed to investigate prognosis and severity of covid-19 infection with using CRP/Albumin ratio in pregnant patient

SUMMARY:
The CRP/albumin ratio (CAR) is a recently defined parameter which represents the ratio of a positive acute phase reactant to a negative acute phase reactant. Recent studies have shown that the CRP/albumin ratio is a biomarker with prognostic value for various inflammatory disorders and serious diseases. With this study it is aimed to investigate the effect of CRP/albumin ratio in predicting the severity and prognosis of the disease in pregnant patients with more severe Covid-19 infection.

DETAILED DESCRIPTION:
Pregnant women are more susceptible to viral infections affecting the respiratory tract than non-pregnant women. Similar to non-pregnant patients, Covid-19 infection occurs with non-specific symptoms in pregnant patients. A computed tomography (CT) scan of lungs and several laboratory parameters are used to predict the prognosis of this infection, which starts with non-specific findings. Although it has been demonstrated that low-dose lung CT can be used safely in pregnant women, both clinicians and pregnant women tend to avoid tomography imaging due to its teratogenic effects

The CRP/albumin ratio (CAR) is a recently defined parameter which represents the ratio of a positive acute phase reactant to a negative acute phase reactant. It is an indicator of both the inflammatory state and the nutritional state, simultaneously. Recent studies have shown that the CRP/albumin ratio is a biomarker with prognostic value for various inflammatory disorders and serious diseases. With this study it is aimed to investigate the effect of CRP/albumin ratio in predicting the severity and prognosis of the disease in pregnant patients with more severe Covid-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Covid PCR test positive patients
* Pregnant

Exclusion Criteria:

* Covid PCR test negative
* Missed data

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: hospitalised Covid PCR test positive pregnant patient
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
CRP/Albumin ratio | First day of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Adıyaman Training and Research Hospital, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No